CLINICAL TRIAL: NCT05688982
Title: MOLAR: Mapping Oral Health and Local Area Resources
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Margaret Samuels-Kalow, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P003224; UH3DE031920 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-05

CONDITIONS: Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A--general information (Other): Patients in Arm A will receive paper handouts with general oral health and aSDoH resources
  Interventions: Behavioral: General information provision
- B--geographic information (Other): Patients in Arm B will receive paper handouts with geographically-proximate oral health and aSDoH resources.
  Interventions: Behavioral: Geographic information provision
- C--geographic information and navigational assistance (Other): Patients in Arm C will receive geographically-proximate oral health and aSDoH resources plus active navigational assistance.
  Interventions: Behavioral: Geographic information provision; Behavioral: Navigational assistance

INTERVENTIONS:
Behavioral: General information provision — Patients will receive information with general oral health and aSDoH resources.
  Arms: A--general information
Behavioral: Geographic information provision — Patients will receive information with geographically-proximate oral health and aSDoH resources based on a directory created by the study team.
  Arms: B--geographic information; C--geographic information and navigational assistance
Behavioral: Navigational assistance — Patients will receive phone-based navigational assistance from the study navigator.
  Arms: C--geographic information and navigational assistance

SUMMARY:
The goal of this clinical trial is to test the impact of a screening and linkage intervention for adverse social determinants of health (aSDoH) on oral health linkage to care for emergency department patients. Researchers will compare three groups: Patients in Arm A will receive paper handouts with general oral health and aSDoH resources. Patients in Arm B will receive paper handouts with geographically-proximate oral health and aSDoH resources. Patients in Arm C will receive geographically-proximate oral health and aSDoH resources plus active navigational assistance.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, an individual must meet all of the following criteria:

  * No evidence of lack of capacity to provide verbal informed consent (as documented in the chart).
  * Willing to comply with all study procedures and be available by phone for the duration of the study (as reported by the patient)
  * Unmet oral health needs as ascertained by the Hope Home (adult) or Gazzaz (pediatric) questions
  * Adult (age ≥18 years old) ED patient or pediatric ED patient (>1 year of age) presenting with parent or legal guardian. Parent will be the primary study participant but if age > 7 years, the child will provide assent for medical record review.
  * Ability to communicate in English or Spanish (as reported by the patient)
  * Emergency severity index (ESI) 2-5 (as documented in the electronic medical record)
  * Residence within catchment area of 3-hospital region (defined by MGB home hospital catchment area) at initial enrollment (as reported by the patient)
  * Working phone number

Exclusion Criteria:

* Patients on involuntary holds (per electronic medical record review)
* Presenting from carceral facilities (per electronic medical record review)
* Presenting for acute mental health care under evaluation for Section 12 (per electronic medical record review)
* Patients presenting for assistance with intimate partner violence (IPV) or care following sexual assault

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2049 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2028-02-22 (Estimated)

PRIMARY OUTCOMES:
Linkage to oral health care | Within 12 months of randomization
  binary, completion of a dental appointment or not

SECONDARY OUTCOMES:
Time to completion of dental appointment at the individual level | Within 12 months of randomization
  continuous, days from randomization to completion of dental appointment
Repeat visits for oral health problems | Within 12 months of randomization
  binary, any return visit or not
Rate of linkage to oral health care at the neighborhood level | Within 12 months of randomization
  continuous rate, ranges from 0-100
Oral health quality of life | Within 12 months of randomization
  Total score on OHIP-14 (continuous, ranges from 0-56) or OHIP-5 (0-20)
Return visits | Within 12 months of initial visit
  Number of return visits to the ED, outpatient visits, inpatient admissions, and ICU admissions (each continuous).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Due to the sensitive nature of the database (including information about potential stigmatizing factors including social risk and need), access to scientific data will be controlled and provided under a restricted data contract to users who demonstrate a valid research need and meet conditions of use. Scientific Data derived from humans will be protected through de-identification, removal of information that may be used to infer the identity of individuals and shared under controlled-access conditions as required by institutional policy.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.

REFERENCES:
- [Derived] Simon L, Marsh R, Sanchez LD, Camargo C, Donoff B, Cardenas V, Manning W, Loo S, Cash RE, Samuels-Kalow ME. Mapping Oral health and Local Area Resources (MOLAR): protocol for a randomised controlled trial connecting emergency department patients with social and dental resources. BMJ Open. 2023 Dec 10;13(12):e078157. doi: 10.1136/bmjopen-2023-078157. PMID 38072485